CLINICAL TRIAL: NCT02746627
Title: Positive Psychology to Improve Adherence in Adolescents With Type 1 Diabetes
Brief Title: Check It! Positive Psychology Intervention to Improve Adherence in Adolescents With T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Jaser, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 131384
Record Dates: First submitted 2016-04-05; First posted 2016-04-21 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants were assigned to Positive Affect - Phone, Positive Affect - Text, or Education groups for the duration of the study.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Education (Active Comparator): Participants receive educational materials in the mail every 2 weeks for 8 weeks.
  Interventions: Behavioral: Education
- Positive Affect - Text (Experimental): Participants receive positive affect intervention (weekly reminders to use gratitude, self-affirmations, parental affirmations, and gift cards) by SMS. Participants also receive educational materials in the mail every 2 weeks for 8 weeks.
  Interventions: Behavioral: Positive Affect; Behavioral: Education
- Positive Affect - Phone (Experimental): Participants receive positive affect intervention (weekly reminders to use gratitude, self-affirmations, parental affirmations) by phone. Participants receive small gifts in the mail every 2 weeks for 8 weeks. educational materials in the mail every 2 weeks for 8 weeks.
  Interventions: Behavioral: Positive Affect; Behavioral: Education

INTERVENTIONS:
Behavioral: Positive Affect — Positive psychology intervention to improve motivation for diabetes management.
  Arms: Positive Affect - Phone; Positive Affect - Text
Behavioral: Education — Educational materials on diabetes management

SUMMARY:
Problems with diabetes management in adolescents with type 1 diabetes are common - occurring at rates as high as 93% - and have serious health consequences, including poor blood sugar control and risk for later complications. Therefore, the investigators proposed to test a positive psychology intervention for adolescents with type 1 diabetes aimed at increasing motivation for diabetes management; specifically, to increase the frequency of blood glucose monitoring. This intervention will boost positive mood in adolescents (age 13-17) through tailored exercises in gratitude, self-affirmation, small gifts, and parent affirmation as a way to improve motivation for diabetes management. In addition, this study will explore the use of technology, by comparing telephone-administered vs. automated text-messaging versions of the intervention, to determine which mode of delivery is more appealing, convenient, and beneficial for adolescents in managing their diabetes.

Participants and parents will complete questionnaires on mood and diabetes management during a routine clinic visits at baseline, 3 months, and 6 months. Clinical measures of diabetes management will be collected from participants' electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes for at least 6 months
* HbA1c between 8-12%
* Speak and read English
* Caregiver living with child

Exclusion Criteria:

* Other uncontrolled health conditions

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savin KL, Hamburger ER, Monzon AD, Patel NJ, Perez KM, Lord JH, Jaser SS. Diabetes-specific family conflict: Informant discrepancies and the impact of parental factors. J Fam Psychol. 2018 Feb;32(1):157-163. doi: 10.1037/fam0000364. PMID 29543490

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone
Started | 60 | 30 | 30
Completed | 59 | 29 | 29
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone | Total
Number analyzed (Participants) | 60 | 29 | 29 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 29 | 29 | 118
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.92 (1.42) | 14.62 (1.63) | 14.97 (1.40) | 14.86 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 12 | 15 | 62
  Male | 25 | 17 | 14 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Non Hispanic | 53 | 26 | 25 | 104
  Black or African american | 2 | 1 | 2 | 5
  Asian | 1 | 0 | 0 | 1
  Biracial/Multiracial | 2 | 0 | 1 | 3
  White Hispanic | 2 | 1 | 1 | 4
  Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 29 | 29 | 118

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control (HbA1c)
Description: HbA1c measured as part of diabetes clinic visit. The target for children and adolescents is <7.5%.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone
Number analyzed (Participants) | 59 | 29 | 29
percentage of glycated hemoglobin | 8.8 [8 to 9.7] | 9 [8.3 to 9.8] | 8.5 [8 to 9]

2. Secondary Outcome: Frequency of Blood Glucose Monitoring
Description: Glucometer download to determine blood glucose checks per day.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: blood glucose checks per day
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone
Number analyzed (Participants) | 49 | 25 | 24
blood glucose checks per day | 3.1 [2.1 to 3.7] | 3.46 [2.6 to 4] | 2.8 [1.9 to 3.51]

3. Secondary Outcome: Diabetes-Related Quality of Life
Description: The Pediatric Quality of Life (PedsQL) Diabetes-Specific Module assesses adolescents' self-reported quality of life. Scaled scores range from 0-100, with higher scores indicating better quality of life.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone
Number analyzed (Participants) | 55 | 25 | 25
score on a scale | 72 [62.5 to 82] | 79 [72 to 82] | 73 [68 to 83]

4. Secondary Outcome: Family Conflict
Description: Diabetes-specific family conflict was measured with the Revised Diabetes Family Conflict Scale, which consists of 19 items regarding how much adolescents and parents argue about diabetes management tasks. Scores range from 19-57, and higher scores indicate greater conflict.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone
Number analyzed (Participants) | 54 | 25 | 25
score on a scale
  Child reported | 23.5 [20 to 36] | 27 [19 to 44] | 36 [21 to 45]
  Parent reported | 23 [22 to 35] | 25 [20 to 29] | 25 [21 to 28]

5. Secondary Outcome: Positive Affect
Description: Positive affect measured using the Positive and Negative Affect Scale for children (PANAS-C). The positive affect scale consists of 15 items. Scores range from 15-75, and higher scores indicate higher levels of positive affect.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone
Number analyzed (Participants) | 59 | 29 | 29
score on a scale | 35 [27.5 to 42.5] | 37 [28 to 42] | 41 [32 to 46]

6. Secondary Outcome: Coping
Description: Responses to Stress Questionnaire measures coping strategies used in response to diabetes-related stress. Scores range from 57-228, and higher scores indicate more responses to stress.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone
Number analyzed (Participants) | 55 | 25 | 25
score on a scale | 107 [91 to 125] | 99 [87 to 126] | 104 [92 to 121]

ADVERSE EVENTS:
Arm/Group | Education | Positive Affect - Text | Positive Affect - Phone
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/60 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No